CLINICAL TRIAL: NCT05313321
Title: Mid-term Survival of the Insignia Stem in Primary Total Hip Arthroplasty
Brief Title: Survival of the Insignia Stem in Total Hip Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lucas Anderson, Principle Investigator, University of Utah
Other Study IDs: 145076
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: Primary Total Hip Arthroplasty; Insignia™ Hip Stem; Radiographic review
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Primary total hip arthroplasty receiving the Insignia Stem: Patients undergoing primary total hip arthroplasty that will likely receive the Insignia Stem and associated Stryker Acetabular Component.
  Interventions: Device: Primary total hip arthroplasty receiving the Insignia Stem

INTERVENTIONS:
Device: Primary total hip arthroplasty receiving the Insignia Stem — Patients receiving the Insignia Stem and associated Stryker Acetabular Component for total hip arthroplasty
  Other Names: Total Hip Arthroplasty

SUMMARY:
The investigators primary objective of this study is to evaluate radiographic fit and fill of the Insignia stem and identify risk factors for aseptic failure. The investigators hypotheses being tested is: the newly designed Insignia stem demonstrates acceptable radiographic fit and fill by reviewing radiolucent lines <2mm.

DETAILED DESCRIPTION:
Total hip arthroplasty is one of the most functionally restorative procedures in modern medicine. Since its introduction in the mid twentieth century significant advancements in implant materials have occurred. There is debate on the design of the femoral stem in total hip arthroplasty. The use of uncemented, Hydroxyapatite (HA)-coated femoral stems have been shown to be reliable and are commonly used. One such implant is the Insignia™ Hip Stem (Stryker, Kalamazoo, MI, USA).

The Insignia™ Hip Stem is a collared stem that features a plasma-sprayed Hydroxyapatite (HA) coating over plasma-sprayed titanium in the proximal region and a plasma-sprayed HA coating over grit blast in the distal region and collar underside. Unfortunately, with it's novelty comes a lack of clinical follow-up and evaluation. As such, the investigators purpose of this study is to evaluate the early radiographic of the Insignia™ Hip Stem.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18
* Patients planning on undergoing primary total hip arthroplasty that will likely receive the Insignia stem and associated Stryker Acetabular Component.
* Preoperative diagnosis of osteoarthritis
* Patients willing and able to comply with follow-up requirements
* Patients willing to sign an IRB approved consent and authorization document

Exclusion Criteria:

* Patients with inflammatory or pyogenic arthritis
* Body Mass Index (BMI)>40
* Bone stock that is inadequate for support or fixation of the prosthesis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning on undergoing primary total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Radiographs review | Pre-operative
  Reviewing radiographic radiolucent lines <2mm
Radiographs review | 6-weeks post-operative
  Reviewing radiographic radiolucent lines <2mm
Radiographs review | 1-year post-operative
  Reviewing radiographic radiolucent lines <2mm
Radiographs review | 2-years post-operative
  Reviewing radiographic radiolucent lines <2mm

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Anderson, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No